CLINICAL TRIAL: NCT06322381
Title: Reinsertion Achilles Tendon VS Zadek Osteotomy in Insertional Achilles Tendinopathy: a Randomized Controlled Trial
Brief Title: Reinsertion Achilles Tendon VS Zadek Osteotomy in Insertional Achilles Tendinopathy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abanoub Henen Helmy Samaan, Resident in Orthopedic department at Assiut university, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Reinsertion AT VS ZO in IAT
Record Dates: First submitted 2024-03-07; First posted 2024-03-21 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Insertional Achilles Tendinopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Reinsertion achilles tendon (Active Comparator): Reinsertion Achilles tendon by 2-4 anchors.
  Interventions: Procedure: Reinsertion achilles tendon
- Zadek osteotomy (Active Comparator): A calcaneal osteotomy was then performed, two Kirschner wires, were then inserted from the posterior aspect of the calcaneus, over which cannulated screws were used for fixation of the osteotomy.
  Interventions: Procedure: Zadek osteotomy

INTERVENTIONS:
Procedure: Reinsertion achilles tendon — Prone position, tourniquet over the thigh, direct midline incision, 2.0 cm proximal the insertion of the Achilles tendon up to 4.0 cm prolonged distal to the insertion is recommended. This is followed by a totally disinsertion of TA. At least a debridement of inflammatory or necrotic tissue as well as the removal of bony tissue is performed. tendon is re-inserted by 2-4 anchors.
  Arms: Reinsertion achilles tendon
Procedure: Zadek osteotomy — lateral position, under spinal anesthesia, tourniquet over the thigh, oblique lateral heel incision starting just anterior to the Achilles tendon, at a 45 angle to the long axis of the calcaneus posterior to the course of the sural nerve. A calcaneal osteotomy was then performed, two Kirschner wires, were then inserted from the posterior aspect of the calcaneus, over which cannulated screws were used for fixation of the osteotomy.
  Arms: Zadek osteotomy

SUMMARY:
The aim of this study is to Compare functional outcome and the recovery time of reinsertion of achilles tendon VS zadek osteotomy in insertional achilles tendinopathy.

DETAILED DESCRIPTION:
Insertional Achilles tendinopathy is characterized by chronic posterior heel pain associated with posterosuperior calcaneal exostosis or intratendinous ossification. The etiologies include retrocalcaneal exostosis, the diseased tendon, enthesopathy, and Haglund's deformity. The nonsurgical therapies, such as physical therapy, stretching and strengthening of the gastrocnemius-soleus muscle complexes, nonsteroid anti-inflammatory drugs, and footwear modifications, are chosen as the initial treatment. Local injection of the steroid is not recommended because it might lead to increase risk of tendon rupture.

Surgical intervention is a suitable option when conservative treatment for more than 6 months has failed. Open detachment with reattachment of the Achilles tendon is a common surgery combined with calcaneoplasty and debridement of the retrocalcaneal bursitis and pathologic Achilles tendon. Suture techniques using bone anchors have been described to reattach the Achilles tendon with excellent results. percutaneous Osteotomy is another option, first described by Zadek in 1939 which was later modified in 1965. zadek osteotomy is a dorsal closing wedge calcaneal osteotomy that allows the tuberosity of Haglund deformity to be brought forward. This operation can change the calcaneus' anatomical length and elevate the distal insertion point of the AT. The rationale of a ZO was to reduce the impingement between the anterior aspect of the Achilles tendon and the superior angle of the posterior calcaneal tuberosity. By shortening the calcaneus and altering the orientation of the Achilles tendon fibers it is believed to decrease stress across the tendon at its insertion.

ELIGIBILITY:
Inclusion Criteria:

* Age range 18 - 65
* Insertional Achilles tendinopathy without steroid injection, infection, tendon rupture and ankle fracture

Exclusion Criteria:

* Age < 18 years, > 65
* General medical contraindications to surgical interventions
* Calcaneal Fracture, subtalar fusion
* infection.
* Pathological tendon rupture
* History of steroid injection

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-02-16 (Estimated); Primary Completion 2025-02-16 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
the time needed to return to normal daily activities (functional outcome) assessed by foot and ankle outcome score. | up to1 year post baseline
  foot and ankle outcome score is a tool to measure the symptoms, stiffness, pain, function, daily living, sports and recreational activities of foot and ankle problems. It is based on 100 questions and ranges from 0 to 100, with higher scores indicating more severe symptoms or limitations.

SECONDARY OUTCOMES:
Pain assessed by the visual analogue scale. | up to1 year post baseline
  The visual analogue scale (VAS) is a scale used to determine the pain intensity experienced by individuals. It consists of a line, approximately 10-15 cm in length, with the left side signifying no pain with a smiling face image and the right side signifying the worst pain ever with a frowning face image. The VAS is used to assist individuals to determine pain levels, who may not be accustomed to rating their pain on other types of scales, such as a numeric rating scale.
Rate of complications | up to1 year post baseline
  Rate of complications e.g. non-union, post-operative infections

CONTACTS AND LOCATIONS:
Overall Officials: Wael Y El-adly, professor, Principal Investigator — Assiut University; Amr AF Mohammed, lecturer, Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Scott A, Huisman E, Khan K. Conservative treatment of chronic Achilles tendinopathy. CMAJ. 2011 Jul 12;183(10):1159-65. doi: 10.1503/cmaj.101680. Epub 2011 Jun 13. No abstract available. PMID 21670110
- [Background] Rees JD, Maffulli N, Cook J. Management of tendinopathy. Am J Sports Med. 2009 Sep;37(9):1855-67. doi: 10.1177/0363546508324283. Epub 2009 Feb 2. PMID 19188560
- [Background] Kleinman M, Gross AE. Achilles tendon rupture following steroid injection. Report of three cases. J Bone Joint Surg Am. 1983 Dec;65(9):1345-7. No abstract available. PMID 6197416
- [Background] Scholten PE, van Dijk CN. Endoscopic calcaneoplasty. Foot Ankle Clin. 2006 Jun;11(2):439-46, viii. doi: 10.1016/j.fcl.2006.02.004. PMID 16798522
- [Background] McAlister JE, Hyer CF. Safety of achilles detachment and reattachment using a standard midline approach to insertional enthesophytes. J Foot Ankle Surg. 2015 Mar-Apr;54(2):214-9. doi: 10.1053/j.jfas.2014.12.009. Epub 2015 Jan 22. PMID 25619811
- [Background] Rigby RB, Cottom JM, Vora A. Early weightbearing using Achilles suture bridge technique for insertional Achilles tendinosis: a review of 43 patients. J Foot Ankle Surg. 2013 Sep-Oct;52(5):575-9. doi: 10.1053/j.jfas.2012.11.004. Epub 2013 May 11. PMID 23669005
- [Background] I. Zadek An operation for the cure of achillobursitis Am J Surg, 43 (1939), pp. 542-546
- [Background] Sanaei-Zadeh H, Emamhadi M, Farajidana H, Zamani N, Amirfarhangi A. Electrocardiographic manifestations in acute methanol poisoning cannot predict mortality. Arh Hig Rada Toksikol. 2013 Jun;64(2):79-85. doi: 10.2478/10004-1254-64-2013-2285. PMID 23819935
- [Background] Georgiannos D, Kitridis D, Bisbinas I. Dorsal closing wedge calcaneal osteotomy for the treatment of Insertional Achilles Tendinopathy: A technical tip to optimize its results and reduce complications. Foot Ankle Surg. 2018 Apr;24(2):115-118. doi: 10.1016/j.fas.2016.12.004. Epub 2016 Dec 30. PMID 29409230